CLINICAL TRIAL: NCT02149303
Title: A Retrospective Cohort Study With Chart Review to Assess the Management of Major Bleeding Events in NVAF Patients Treated With Dabigatran Etexilate
Brief Title: Management of Major Bleeding Events in Atrial Fibrillation Patients Using Pradaxa
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.200
Record Dates: First submitted 2014-05-19; First posted 2014-05-29 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Atrial Fibrillation; Hemorrhage
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Dabigatran
  Interventions: Drug: Dabigatran 75 mg; Drug: Dabigatran 150 mg

INTERVENTIONS:
Drug: Dabigatran 75 mg — PO BID
Drug: Dabigatran 150 mg — PO BID

SUMMARY:
This study is being conducted to collect data on the management of major bleeding events occurring in patients with atrial fibrillation taking dabigatran etexilate.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* Greater than or equal to 18 years of age;
* Confirmed diagnosis of non valvular atrial fibrillation (NVAF) (Diagnosis of AF is considered confirmed if there is medical chart documentation that the patient has atrial fibrillation or AF or the ICD-9 or ICD-10 code for AF is documented);
* NVAF is defined as follows: nonvalvular atrial fibrillation is restricted to cases in which the rhythm disturbance occurs in the absence of rheumatic mitral stenosis or a prosthetic heart valve.
* Documentation that the patient presented to an emergency department/emergency room (ED/ER) for a major bleeding event (index event);
* Major bleeding is defined by International Society on Thrombosis and Haemostasis (ISTH) as:
* fatal bleeding and/or
* symptomatic bleeding in a critical area/organ such as intracranial, intraspinal, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular with compartment syndrome, and/or
* bleeding causing a fall in hemoglobin of 20g per liter or more, or leading to transfusion of 2 or more units of whole blood or red blood cells
* Documentation that the index event occurred in a patient who reported having taken at least one dose of dabigatran within the 5 days prior to the index event.

Exclusion criteria:

* Confirmed diagnosis of valvular AF (Diagnosis of valvular AF is considered confirmed if there is medical chart documentation that the patient has valvular AF or VAF. In the absence of documentation to indicate whether the patient has non-valvular or valvular AF,);
* Documentation that the patient was taking dabigatran with a concomitant anticoagulant (contemporaneous parenteral anticoagulant or another oral anticoagulant) within 72 hours of the index event;
* The concomitant administration of antiplatelet medications prior to the onset of the index event is not exclusionary;
* Documentation of the patient receiving thrombolytic therapy within 48 hours of the onset of the index event;
* Documentation that the patient was enrolled in an interventional investigational or other BI observational clinical trial at the time of the onset of the index event;
* Medical record was not retrievable, was missing or empty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AF patients with bleeding event using Dabigatran etexilate
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- United States (5):
  - 1160.200.02 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1160.200.06 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1160.200.01 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 1160.200.05 Boehringer Ingelheim Investigational Site, Stony Brook, New York
  - 1160.200.03 Boehringer Ingelheim Investigational Site, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a retrospective observational study. 284 subjects were captured in the initial screening. 93 subjects were found not to meet the eligibility criteria and were excluded from the study, leaving 191 subjects eligible for study entry who were enrolled and included in the final study.
Groups:
- Dabigatran Etexilate (Pradaxa®): Patients with Non-Valvular Atrial Fibrillation (NVAF) at five U.S. sites who received dabigatran (at the 75 mg and 150 mg dosages, orally twice daily), who had an acute bleeding event (index event), and either presented to an Emergency Department/ Emergency Room (ED / ER) or were hospitalized primarily for management of a major bleeding event.
Period: Overall Study
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Started | 191
Completed | 191
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who received treatment at the five study sites.
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.6 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 98

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Index Event Safety Outcomes (Resolved / Recovery Ongoing / Deceased) at the Time of Their Hospital Discharge / Release.
Description: Proportion of subjects with index event safety outcomes (resolved / recovery ongoing / deceased) at the time of their hospital discharge / release.
Time Frame: From the time of presentation / admission to an ED / ER or hospitalization through all in-hospital referrals until discharge (between 20 August 2014 (the date of the first data entry) and 4 March 2015 (the date of data entry closure)); Up to 196 days
Population: Patients who received treatment at the five study sites
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 191
Percentage of participants
  Resolved at discharge | 86.4
  Unresolved at discharge (Recovery ongoing) | 7.3
  Died before discharge (Deceased) | 6.3

2. Primary Outcome: Proportion of Subjects Receiving Different Types of Interventions (i.e., Medication / Procedure and Surgery) to Manage the Index Events Until Their Hospital Discharge / Release
Description: Proportion of subjects receiving different types of interventions (i.e., medication / procedure and surgery) to manage the index events until their hospital discharge / release.
Time Frame: as for outcome 1
Population: Patients who received treatment at the five study sites
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 191
Percentage of participants
  Fluid transfusion | 72.8
  Blood transfusion | 57.1
  Fresh frozen plasma (FFP) | 24.6
  Plasma cryoprecipitate | 1.6
  Platelets | 5.8
  Blood coagulation factor concentrates | 5.8
  Computed tomography (CT) scanning | 39.3
  X-ray | 24.1
  Upper endoscopy | 20.9
  Colonoscopy | 19.9
  Endoscopy (unspecified whether lower or upper) | 6.3
  Nuclear imaging | 5.8
  Ultrasound | 5.8
  Magnetic resonance imaging (MRI) | 3.7
  Enteroscopy | 1.6
  Sigmoidoscopy | 1.6
  Surgery or procedure | 26.7
  Drugs for the alimentary tract | 32.5
  Blood/anticoagulant medication | 7.9
  Vitamin K | 3.7

3. Primary Outcome: Index Event Characteristics (i.e. Type of Bleeding and Anatomic Locations of the Index Event) at the Time of the ED / ER Presentation or Hospitalization
Description: Proportion of Index events by anatomic location and type are presented. The categories of Unknown and Other presented below correspond to, Unknown: Unknown location of bleeding met the criteria for major bleeding as defined by the International Society on Thrombosis and Haemostasis (ISTH).
  Other: Other types of bleeding represent a combined category of all other locations of bleeding whose incidence was <1.7%.
Time Frame: as for outcome 1
Population: Patients who received treatment at the five study sites
Measure: Number; unit: Percentage of events
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Number analyzed (Participants) | 191
Percentage of events
  Gastrointestinal | 61.8
  Upper tract | 22.5
  Lower tract | 34.0
  Brain / Intracranial | 18.8
  Non-trauma | 4.2
  Trauma | 14.7
  Fall | 14.1
  Motor vehicle accident | 0.5
  Unknown | 0.5
  Other | 18.8

ADVERSE EVENTS:
Time Frame: From the time of presentation / admission to an ED / ER or hospitalization through all in-hospital referrals until discharge (between 20 August 2014 (the date of the first data entry) and 4 March 2015 (the date of data entry closure)); Up to 196 days
Arm/Group | Dabigatran Etexilate (Pradaxa®)
Serious Adverse Events (participants affected / at risk) | 11/191
Other Adverse Events (participants affected / at risk) | 50/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (Pradaxa®) (N=191)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate (Pradaxa®) (N=191)
Anaemia (Blood and lymphatic system disorders) | 34
Diverticulum (Gastrointestinal disorders) | 14
Haemorrhoids (Gastrointestinal disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights